CLINICAL TRIAL: NCT04132466
Title: ASSURE WCD Clinical Evaluation - Conversion Efficacy Study (ACE-CONVERT)
Brief Title: ASSURE WCD Clinical Evaluation - Conversion Efficacy Study
Acronym: ACE-CONVERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kestra Medical Technologies, Inc. (Industry)
Collaborators: Regulatory and Clinical Research Institute Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3333934_C
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Death, Sudden, Cardiac
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: Multicenter single arm open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Enrolled Subjects (Experimental): Adult subjects who met eligibility criteria and provided written informed consent to participate
  Interventions: Device: Defibrillation using the ASSURE wearable cardioverter defibrillator therapy delivered via a waveform delivery test system

INTERVENTIONS:
Device: Defibrillation using the ASSURE wearable cardioverter defibrillator therapy delivered via a waveform delivery test system — defibrillation using a 170 joule biphasic truncated exponential waveform designed for the ASSURE wearable cardioverter defibrillator

SUMMARY:
A multicenter single arm open label evaluation of the ASSURE Wearable Cardioverter Defibrillator (WCD) defibrillation waveform in adult cardiac patients

DETAILED DESCRIPTION:
The objective of this study is to evaluate Ventricular Tachycardia/Ventricular Fibrillation (VT/VF) conversion efficacy in adult human subjects using the ASSURE Wearable Cardioverter Defibrillator (WCD) defibrillation waveform.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age ≥ 18 years
2. Able and willing to provide written informed consent before undergoing any study-related procedures
3. Scheduled for any of the following procedures:

   1. Electrophysiology study for induction of ventricular arrhythmias
   2. Non-invasive electrophysiology testing using an existing implantable defibrillator
   3. Implantable cardioverter-defibrillator (ICD) replacement procedure during which induction of a ventricular arrhythmia is planned
   4. Ablation of ventricular tachycardia (patients undergoing ventricular tachycardia ablation in which only a substrate modification approach is planned, with no intention of inducing a ventricular arrhythmia, should not be included)

Exclusion Criteria:

1. Any condition that by the judgement of the physician investigator precludes the subject's ability to comply with the study requirements
2. Pregnancy
3. Use of mechanical circulatory support (e.g. Left Ventricular Assist Device, Total Artificial Heart, intraaortic balloon pump or Impella)
4. Documented nonchronic cardiac thrombus
5. Atrial fibrillation or atrial flutter without therapeutic systemic anticoagulation
6. Critical aortic stenosis
7. Unstable coronary artery disease (CAD)
8. Recent stroke or transient ischemic attack (TIA)
9. Hemodynamic instability
10. Currently implanted Boston Scientific S-ICD (due to location of implant relative to test system)
11. Unstable angina
12. New York Heart Association (NYHA) Class IV
13. Left Ventricular Ejection Fraction (LVEF) < 20%
14. Any medical condition that by the judgement of the physician investigator, patient participation in this study is not in the best interest of the patient
15. History of difficulty of ventricular arrhythmia induction
16. Amiodarone use within 3 months before the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marye Gleva, MD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Alaska Cardiovascular Research Foundation, Inc., Anchorage, Alaska
  - University of Michigan, Ann Arbor, Michigan
  - Washington University St Louis, St Louis, Missouri
  - Institute for Research and Innovation MultiCare Health System, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gleva MJ, Sullivan J, Crawford TC, Walcott G, Birgersdotter-Green U, Branch KR, Doshi RN, Kivilaid K, Brennan K, Rowbotham RK, Gustavson LM, Poole JE. Defibrillation effectiveness and safety of the shock waveform used in a contemporary wearable cardioverter defibrillator: Results from animal and human studies. PLoS One. 2023 Mar 14;18(3):e0281340. doi: 10.1371/journal.pone.0281340. eCollection 2023. PMID 36917566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen (13) patients were enrolled at two investigational sites between November 25, 2019 and March 19, 2020. In consult with the FDA, enrollment was stopped short of the target enrollment of 20 patients due to the COVID-19 outbreak.
Period: Overall Study
Arm/Group | Enrolled Subjects
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Cumulative First and Second Shock VT/VF Conversion Rate
Description: The number of subjects with successful (first or second shock) arrhythmia conversion using the Test System divided by the total number of inductions attempted using the Test System
  A successful arrhythmia conversion is defined as termination of an induced ventricular rhythm by first or second shock from the Test System to a non-shockable rhythm (rhythms other than VT or VF).
Time Frame: Through study procedure completion, average of 2 hours
Population: In consult with FDA, enrollment was halted due to the COVID pandemic after 13 subjects were enrolled. The study procedure was completed on all 13 subjects, which comprised the Intention-to-Treat cohort. Study monitoring identified one subject had been prescribed Amiodarone during an emergency room visit (three weeks prior to study enrollment) and continued taking it for 6 days (protocol eligibility deviation). Twelve patients were therefore included in the Per Protocol cohort.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Per-Protocol: Adult subjects who met eligibility criteria and provided written informed consent to participate
  Defibrillation using the ASSURE wearable cardioverter defibrillator therapy delivered via a waveform delivery test system: defibrillation using a 170 joule biphasic truncated exponential waveform designed for the ASSURE wearable cardioverter defibrillator
- Intention-to-Treat: All subjects enrolled
Arm/Group | Per-Protocol | Intention-to-Treat
Number analyzed (Participants) | 12 | 13
percentage | 100 [73.5 to 100] | 100 [75.3 to 100]

2. Secondary Outcome: First Shock VT/VF Conversion Rate
Description: The number of subjects with successful (first shock) arrhythmia conversion using the Test System divided by the total number of inductions attempted with using the Test System
  A successful arrhythmia conversion is defined as termination of an induced ventricular rhythm by first shock from the Test System to a non-shockable rhythm (rhythms other than VT or VF).
Time Frame: Through study procedure completion, average of 2 hours
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Per-Protocol | Intention-to-Treat
Number analyzed (Participants) | 12 | 13
percentage | 83.3 [51.6 to 97.9] | 84.6 [54.6 to 98.1]

ADVERSE EVENTS:
Time Frame: During the study procedure or observed during clinical follow-up within one week post procedure.
Description: Adverse events in this study were limited to adverse device effects (ADEs). An ADE was defined as any untoward medical occurrence in a subject during the study that in the opinion of the investigator is at least possibly related to use of the Test System during the study procedure. Anticipated adverse device effects were specified in the study protocol based on risk assessment.
Arm/Group | Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=13)
Redness/Irritation (Anticipated Adverse Device Effect) (Skin and subcutaneous tissue disorders) | 3 (3) — Mild skin irritation and redness in the location of the defibrillation pads within 48 hours following the procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04132466/Prot_SAP_000.pdf